CLINICAL TRIAL: NCT04776707
Title: Investigation of the Validity and Reliability of the Turkish Translation of the Sensory Hypersensitivity Scale
Brief Title: Reliability and Validity of the Turkish Version of Sensory Hypersensivity Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.115
Record Dates: First submitted 2021-02-19; First posted 2021-03-02 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-01

CONDITIONS: Central Sensitisation; Hypersensitivity
Keywords: central sensitization; chronic pain; sensory hypersensitivity; Sensory hypersensitivity scale; Central sensitization inventory
MeSH Terms: conditions — Hypersensitivity; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Central sensitization (CS) is as increased response to normal or sub-threshold stimuli of central nervous system. Patient history and physical examination, quantitative sensory testing(QST), imaging methods, neuroinflammatory marker levels, electrodiagnostic studies and clinical scales can be used in the diagnosis of CS, but there is no standardized method yet. Among these methods, clinical scales are preferred because they are practical, inexpensive and do not require experience. The Sensory Hypersensitivity Scale was developed by Dixon et al. for investigate the personal hypersensitivity and CS. The aim of this study is to investigate the Turkish validity and reliability of the sensory hypersensitivity scale.

DETAILED DESCRIPTION:
The term central sensitization (CS) was first used by Wolf in 1988 and was explained as the increase in pain sensitivity with the amplification of neuron-derived signals in the central nervous system. With the development of CS, a decrease in the pain threshold and an increase in generalized sensitivity occur. There is no method for the diagnosis of CS is accepted as a gold standard. Clinical scales and quantitative sensory testing (QST) is used for this purpose widely. In addition, the well-known scale used for the evaluation of CS is the Central Sensitization Inventory (CSI), developed for detect CS in chronic pain patients. The use of CSI, which is more practical to use, is becoming widespread because QST takes time, is costly and requires experienced practitioners. Considering the place of sensory hypersensitivity in the diagnosis of CS and the application difficulties of QST, the Sensory Hypersensitivity Scale was developed in 2016. This scale includes 25 questions in the form of a Likert scale and questions the increase in modality-specific (touch, taste, hearing, etc.) sensitivity as well as the general sensitivity increase. Especially in chronic pain conditions, there is an increase in the evidence regarding the development of CS day by day, and the need for auxiliary tools in diagnosis is increasing in parallel. In this study, it was planned to show the Turkish reliability and validity the Sensory Hypersensitivity Scale.

ELIGIBILITY:
Inclusion Criteria:

* Have musculoskeletal pain that lasts for at least 3 months
* Accepting to participate in the study

Exclusion Criteria:

* Refuse to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients aged 18-75 years diagnosed with chronic musculoskeletal disorders will be recruited from a PMR outpatient clinic of a state hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-16 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Sensory hypersensitivity scale | 6 months
  Standardized questionnaire to detective sensor hypersensitivity. This scale includes 25 questions in the form of a Likert scale and questions the increase in modality-specific (touch, taste, hearing, etc.) sensitivity as well as the general sensitivity increase. It is accepted that the higher the score, the higher the sensory hypersensitivity.
Central sensitization inventory | 6 months
  25 somatic and psychosocial symptoms, which are frequently found in patients with central sensitization in part A, are questioned. In part B, the presence of diseases whose relationship with central sensitization is well defined is questioned in the patient without participating in scoring. Central sensitization is assumed in patients who score 40 or more over 100 points.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  This scale included the 14 item checklist in which 7 items relate to anxiety. A subscore of > 8 for depression or anxiety would indicate a clinical case.

SECONDARY OUTCOMES:
VAS pain | 6 months
  The patients pain severity will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Canan ŞANAL TOPRAK, Asst.Prof, Study Chair — Marmara University
Locations (1):
- Feyza Nur YUCEL, Sinop, Boyabat, Turkey (Türkiye)

REFERENCES:
- [Background] Woolf CJ, Thompson SW, King AE. Prolonged primary afferent induced alterations in dorsal horn neurones, an intracellular analysis in vivo and in vitro. J Physiol (Paris). 1988-1989;83(3):255-66. PMID 3272296
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Dixon EA, Benham G, Sturgeon JA, Mackey S, Johnson KA, Younger J. Development of the Sensory Hypersensitivity Scale (SHS): a self-report tool for assessing sensitivity to sensory stimuli. J Behav Med. 2016 Jun;39(3):537-50. doi: 10.1007/s10865-016-9720-3. Epub 2016 Feb 12. PMID 26873609
- [Background] Maguire M. The psychopharmacology of epilepsy. Handb Clin Neurol. 2019;165:207-227. doi: 10.1016/B978-0-444-64012-3.00012-5. PMID 31727213